CLINICAL TRIAL: NCT04625010
Title: The Effectiveness of Two Different Methods Applied During Heel Blood Collection on Pain Level of Healthy Term Newborns
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Collaborators: Bandırma Onyedi Eylül University (Other)
Responsible Party: Principal Investigator, Sevil Inal, Prof. Dr., Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IstanbullUC
Record Dates: First submitted 2020-11-06; First posted 2020-11-12 (Actual); Last update posted 2020-11-12 (Actual); Status verified 2020-11

CONDITIONS: Newborn; Pain; Maternal; Procedure; Needle Stick
Keywords: Newborn; Pain management; Swaddling; Maternal holding; Heel stick
MeSH Terms: conditions — Pain; Needlestick Injuries; Agnosia

STUDY DESIGN:
Intervention Model Description: Prospective, randomized controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group 2 (Swaddling group) (Experimental): Swaddling group: Swaddling is a wrapping procedure in which a baby's arms and legs are comfortable, sometimes only the arms are wrapped inside, and two ends of fabric are crossed on the chest of the baby, generally with thin cotton and soft fabric or a blanket. In the swaddling group, neonates were placed in the supine position on a blanket. In compliance with the newborn anatomic posture, the legs were wrapped in the flexion and abduction position. The arms of the neonates were placed close to their torso with both hands, without restraining limb movements. Swaddling was carried out 1 minute before the heel stich procedure and continued 3 minutes after the procedure. The neonate remained on the examination table during the swaddling procedure. Swaddling was applied not too loose or too tight during the procedure.
  Interventions: Other: Swaddling
- Group 3 (Maternal Holding group) (Experimental): Maternal holding group: Neonates in this group were held in their mothers' lap while their mothers were seated reclining on a comfortable chair. Neonates remained clothed in their mothers' lap during the heel stick procedure, and no breastfeeding was administered during the procedure. Holding was continued for a minimum of 3 minutes during and after the procedure.
  Interventions: Other: Maternal holding
- Group 1 (No Intervention): In the control group, the heel stick procedures were conducted using the standard method and the neonates received no interventions during the procedures.

INTERVENTIONS:
Other: Swaddling — Swaddling is a wrapping procedure in which a baby's arms and legs are comfortable, sometimes only the arms are wrapped inside, and two ends of fabric are crossed on the chest of the baby, generally with thin cotton and soft fabric or a blanket. In the swaddling group, neonates were placed in the supine position on a blanket. In compliance with the newborn anatomic posture, the legs were wrapped in the flexion and abduction position. The arms of the neonates were placed close to their torso with both hands, without restraining limb movements. Swaddling was carried out 1 minute before the heel stich procedure and continued 3 minutes after the procedure. The neonate remained on the examination table during the swaddling procedure. Swaddling was applied not too loose or too tight during the procedure.
  Other Names: Group 2
  Arms: Group 2 (Swaddling group)
Other: Maternal holding — Neonates in this group were held in their mothers' lap while their mothers were seated reclining on a comfortable chair. Neonates remained clothed in their mothers' lap during the heel stick procedure, and no breastfeeding was administered during the procedure. Holding was continued for a minimum of 3 minutes during and after the procedure.
  Other Names: Group 3
  Arms: Group 3 (Maternal Holding group)

SUMMARY:
This study was planned to evaluate the effect of two different non-pharmacologic pain relief methods (swaddling and maternal holding) on healthy term newborn's pain levels during heel stick.

Study hypotheses are; Hypothesis 1. Swaddling is effective at relieving pain due to heel stick procedures in newborns. Hypothesis 2. Maternal holding is effective at relieving pain due to heel stick in newborns. Hypothesis 3. Maternal holding is more effective than swaddling at relieving pain due to heel stick in newborns.

DETAILED DESCRIPTION:
This study was conducted in the baby's nursery of Bandirma State Hospital, Turkey between March and June 2016. It was designed as a prospective randomized clinical trial that evaluated and experimentally determined the effects of swaddling and maternal holding during heel stick on pain levels in healthy term neonates.

The study comprised all newborns who came to the baby's nursery for a heel stick procedure for routine metabolic screening; the study sample consisted of 105 healthy newborns who matched the case selection criteria and underwent heel stick. The inclusion criteria were as follows: full term neonates (38-42 weeks of gestation) who underwent heel stick blood drawing for routine metabolic screening, were aged 2 to 4 days, and had passed the hearing screening. Babies with congenital anomalies were excluded from the study.

In the power analysis conducted using heel stick literature1,4,9, the sample size required for 80% reliability and α=0.05 was 35 in each group; the total was 105. Neonates were randomized into three groups and 35 babies were evaluated in each group (swaddling [n=35], maternal holding [n=35], control [n=35]) (Figure 1). Numbers from 1-105 were randomly distributed by a computer program to the three groups with no number repetition to determine which child would be allocated to which group.

The study data were obtained using an information form and the Neonatal Infant Pain Scale (NIPS).

Information Form: This form contained questions about the sociodemographic characteristics of the neonate and family. It consisted of 20 questions in total comprising personal characteristics information of the families, and sex, delivery method (vaginal or cesarean), gestational age, birth weight, postnatal age (hours after birth) of the neonate and period of procedures.

Neonatal Infant Pain Scale: NIPS was developed by Lawrence et al. (1993)21 to evaluate behavioral and physiologic pain responses of preterm and term infants. The scale was adapted to Turkish by Akdovan (1999)22. In the present study, NIPS was used to evaluate the interventional (procedural) pain level of newborns. The scale consists of five behavioral (facial expressions, crying, wakefulness, arm and leg movements) and a physiologic (breathing) signs; 0-2 points are given to the crying indicator, 0-1 points are given to other indicators, and the total score is between 0 and 7. High scores indicate that the severity of pain is excessive.

Data collection All blood sampling was performed in a quiet nursery room between 09:00 AM and 11:00 AM, 1-2 hours after breastfeeding, the normal time when infants undergo heel stick for routine blood collection for metabolic screening. Blood collection was performed in a standardized manner by the same nurse who has a minimum of 5 years' experience in the performance heel stick and had no conflict of interest. A pediatrician made the clinical decision for heel stick.

Before the procedure, the newborns were kept in a quiet room far away from the cries of other babies. The infants' diapers were changed before procedure. For the heel stick procedure, the antiseptic solution (70% alcohol), heel stick method, heel region for sampling (the outer right side of the ball), needle (21-G needle), and environmental factors such as heat, light, and noise were all standardized. The whole procedure was video-recorded until three minutes after the procedure.

At the beginning of the study, the parents of the newborns were informed about the aim and content of the research, and parental approval was obtained. Neonatal and family demographics were collected using self-report information forms, which included medical history, mother's gestational age, neonatal age, sex, birth weight, duration of sampling, total crying time, processing time, and the time from the start of the first cry to the first crying during the process.

All blood sampling in the study was performed for clinical purposes, such as newborn metabolic screening tests, which were taken on the second to third days following birth. The standard protocol for blood sampling involved swabbing the heel with a small gauze pad with disinfectant, lancing the heel, and then gently squeezing the heel intermittently until the amount of blood required for clinical use was collected.

All procedures performed in the experimental and control groups were video recorded by the researcher from the beginning of the procedure. After the procedure the newborns' pain levels and crying duration were evaluated using the video recordings. Assessment of pain was conducted independently by the investigator and the nurse using NIPS. At the same time, the newborns' total procedural crying time, the duration of the procedure, and the first calming time were recorded. The total crying time of the newborns was measured from the start of crying due to heel stick to the complete cessation of crying. The time of the procedure was measured from the beginning to the end of the heel stick procedure. The calming time was measured from the time of the first cry to the first calming time.

The SPSS (version 19) program was used for statistical analysis. Descriptive statistical methods (mean, standard deviation, median, frequency, rate, min., max.) were used when study data were evaluated. The one-way Anova test was used in the comparison of data of the three groups with normal distribution. The Kruskal-Wallis test was used in the comparison of data of the three groups with non-normal distribution. The Mann-Whitney U test was used to identify the group that caused the difference. Pearson's Chi-square test and the Fisher-Freeman-Halton test were used for the comparison of qualitative data. Significance was considered as p<0.05.

ELIGIBILITY:
Inclusion Criteria:

* full term neonates (38-42 weeks of gestation)
* underwent heel stick blood drawing for routine metabolic screening,
* aged 2 to 4 days
* passed the hearing screening

Exclusion Criteria:

* Congenital anomalies

Ages: 2 Days to 4 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 105 (Actual)
Dates: Start 2016-03-01 (Actual); Primary Completion 2016-06-01 (Actual); Study Completion 2016-12-30 (Actual)

PRIMARY OUTCOMES:
NIPS (Neonatal Infant Pain Scale) | Pain levels of the newborns evaluated during the procedures
  Neonatal Infant Pain Scale: NIPS was developed by Lawrence et al. (1993)21 to evaluate behavioral and physiologic pain responses of preterm and term infants. The scale was adapted to Turkish by Akdovan (1999)22. In the present study, NIPS was used to evaluate the interventional (procedural) pain level of newborns. The scale consists of five behavioral (facial expressions, crying, wakefulness, arm and leg movements) and a physiologic (breathing) signs; 0-2 points are given to the crying indicator, 0-1 points are given to other indicators, and the total score is between 0 and 7. High scores indicate that the severity of pain is excessive.

SECONDARY OUTCOMES:
Total criying time | The time of the procedure was measured from the beginning to the end of the heel stick procedure.
  The total crying time of the newborns was measured from the start of crying due to heel stick to the complete cessation of crying.
The time to first calming | Procedure (The calming time was measured from the time of the first cry to the first calming time.)
  The calming time was measured from the time of the first cry to the first calming time.

CONTACTS AND LOCATIONS:
Overall Officials: Leyla Erdim, Dr, Principal Investigator — Istanbul University - Cerrahpasa
Locations (1):
- Sevil İnal, Istanbul, Büyükçekmece, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
I did not find It appropriate to share it.

REFERENCES:
- [Background] Gradin M, Eriksson M, Holmqvist G, Holstein A, Schollin J. Pain reduction at venipuncture in newborns: oral glucose compared with local anesthetic cream. Pediatrics. 2002 Dec;110(6):1053-7. doi: 10.1542/peds.110.6.1053. PMID 12456899
- [Result] Obeidat HM, Shuriquie MA. Effect of Breast-Feeding and Maternal Holding in Relieving Painful Responses in Full-Term Neonates: A Randomized Clinical Trial. J Perinat Neonatal Nurs. 2015 Jul-Sep;29(3):248-54. doi: 10.1097/JPN.0000000000000121. PMID 26218818
- [Result] Okan F, Ozdil A, Bulbul A, Yapici Z, Nuhoglu A. Analgesic effects of skin-to-skin contact and breastfeeding in procedural pain in healthy term neonates. Ann Trop Paediatr. 2010;30(2):119-28. doi: 10.1179/146532810X12703902516121. PMID 20522298
- [Result] Harrison D, Reszel J, Bueno M, Sampson M, Shah VS, Taddio A, Larocque C, Turner L. Breastfeeding for procedural pain in infants beyond the neonatal period. Cochrane Database Syst Rev. 2016 Oct 28;10(10):CD011248. doi: 10.1002/14651858.CD011248.pub2. PMID 27792244
- [Result] Karakoc A, Turker F. Effects of white noise and holding on pain perception in newborns. Pain Manag Nurs. 2014 Dec;15(4):864-70. doi: 10.1016/j.pmn.2014.01.002. Epub 2014 Feb 20. PMID 24559599
- [Result] Morrow C, Hidinger A, Wilkinson-Faulk D. Reducing neonatal pain during routine heel lance procedures. MCN Am J Matern Child Nurs. 2010 Nov-Dec;35(6):346-54; quiz 354-6. doi: 10.1097/NMC.0b013e3181f4fc53. PMID 20926970
- [Result] Cong X. Heel stick test for obtaining blood samples in neonates: both swaddling and heel warming may help, but heel warming appears to provide greater pain reduction. Evid Based Nurs. 2015 Oct;18(4):118. doi: 10.1136/eb-2014-102048. Epub 2015 Apr 16. No abstract available. PMID 25883132